CLINICAL TRIAL: NCT05328804
Title: Evaluating the Efficacy and Safety of the Combination of Herombopag and Human Thrombopoietin (rhTPO) in the Treatment of Patients With Severe Immune Thrombocytopenia (ITP)
Brief Title: Herombopag + rhTPO in Severe Immune Thrombocytopenia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yin Jie (Other)
Responsible Party: Sponsor-Investigator, Yin Jie, Physician, The First Affiliated Hospital of Soochow University
Organization: The First Affiliated Hospital of Soochow University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ-ITP01
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Immune Thrombocytopenia
Keywords: immune thrombocytopenia; severe; Herombopag; recombinant human thrombopoietin
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Patients with severe ITP will be randomly assigned to three groups: rhTPO group, Herombopag Group, Herombopag combined with rhTPO group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- rhTPO (Experimental): rhTPO will be injected subcutaneously at 300 u/kg daily for 14 days.
  Interventions: Drug: rhTPO
- Herombopag (Experimental): Herombopag will be taken orally at 5 mg daily for 28 days.
  Interventions: Drug: Herombopag
- Herombopag in combination of rhTPO (Experimental): Herombopag will be taken orally at 5 mg daily for 28 days，while rhTPO will be injected subcutaneously at 300 u/kg daily for 14 days
  Interventions: Drug: rhTPO; Drug: Herombopag

INTERVENTIONS:
Drug: rhTPO — subcutaneous injection
  Arms: Herombopag in combination of rhTPO; rhTPO
Drug: Herombopag — Orally by mouth
  Arms: Herombopag; Herombopag in combination of rhTPO

SUMMARY:
Severe immune thrombocytopenia (ITP) is a life-threatening acquired hemorrhagic disease with dramatically decreased platelet number and clinical bleeding symptoms. Some patients with severe ITP did not respond to first-line treatment including steroids and IVIG. It was critical for them to use effective treatments to promote platelet and reduce the risk of fatal bleeding. In this study, the patients with severe ITP will be treated with hetrombopag, rhTPO, and the combination of hetrombopag and rhTPO, respectively. The effect evaluation includes the increase of platelet number and decrease of bleeding scores. Changes of coagulation, platelet activation, fribrinolysis influence, and thrombotic events will also be accessed for the safety of treatments. The aim of this study is to demonstrate that the combination of hetrombopag and rhTPO for severe ITP is more effective than the other two monotherapy and does not increase thrombotic events or thrombosis risk.

DETAILED DESCRIPTION:
Patients with severe ITP will be randomly assigned to three groups: rhTPO group, Herombopag Group, Herombopag combined with rhTPO group. The effective rate of treatment, the rate and amplitude of platelet increase, the response time of platelet maintenance, and the effect of combination therapy on hemostasis will be compared. At the same time, the investigators will analyze the markers of thrombosis and thrombotic events to assess the safety of combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female,70 ≥age≥18；
2. Diagnosed as primary immune thrombocytopenia；
3. Platelet count was less than 10 × 10E9 / L with active bleeding, or bleeding score ≥ 5 points；
4. No use of IVIG, Avatrombopag, Eltrombopag or Romiplostim 2 weeks before treatment；
5. Rituximab was used for at least 2 months, and other immunosuppressants were stable for at least 4 weeks.
6. There was no history of platelet transfusion one week before treatment.

Exclusion Criteria:

1. Secondary thrombocytopenia caused by other autoimmune diseases and virus infection was excluded；
2. Patients with active malignant tumors, pregnancy, severe cardiovascular， cerebrovascular diseases and a history of arteriovenous thrombotic diseases were excluded；
3. Patients deemed unsuitable for enrollment by the investigator；
4. Patients with thrombotic disease or serious uncontrolled cardiovascular and cerebrovascular disease;
5. Patients reject to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | From randomization to 28 days after rhTPO/Herombopag/Herombopag+rhTPO treatment
  platelets ≥30*10E9/L, and at least 2 times higher than the baseline platelet count, and there is no hemorrhagic manifestations
The rate and magnitude of the increase in platelet count | From randomization to 28 days after rhTPO/Herombopag/Herombopag+rhTPO treatment
  The rate and magnitude of the increase in platelet count after treatment
Platelet maintenance response time | From randomization to 28 days after rhTPO/Herombopag/Herombopag+rhTPO treatment
  Platelets stay above 30*10E9/L

SECONDARY OUTCOMES:
Platelet fuction | From randomization to 28 days after rhTPO/Herombopag/Herombopag+rhTPO treatment
  Platelet aggregation function assay and the expression of P selectin on platelet surface
the markers of thrombosis and fibrinolysis | From randomization to 28 days after rhTPO/Herombopag/Herombopag+rhTPO treatment
  platelet-derived microparticals in plasma, concentration of Plasminogen Activator Inhibitor-1 （PAI-1）, D-D dimer, tissue plasminogen activator （tPA），urokinase-type plasminogen activator （uPA） and Thrombin activatable fibrinolysis inhibitor （TAFI）
Thrombotic events | From randomization to 3 months after rhTPO/Herombopag/Herombopag+rhTPO treatment
  the number/time/site of thrombotic events （lower extremity deep vein thrombosis, pulmonary embolism, intracranial thrombosis, .etc）in participants

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yin, Principal Investigator — First Affiliated Hospital of Soochow University
Locations (1):
- Jie Yin, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No